CLINICAL TRIAL: NCT05726279
Title: PROtecting Maternal Brains From Injury and Stroke (PROMIS)
Brief Title: PROtecting Maternal Brains From Injury and Stroke
Acronym: PROMIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Randolph S. Marshall, MD, Professor of Neurology, Columbia University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AAAU3179; 5R21HD110992-02 (NIH)
Record Dates: First submitted 2023-02-03; First posted 2023-02-13 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Preeclampsia; Maternal Hypertension
Keywords: Pregnancy; Near-Infrared Spectroscopy (NIRS); Preeclampsia; Maternal health
MeSH Terms: conditions — Pre-Eclampsia; Hypertension, Pregnancy-Induced

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Observational Cohort (No Intervention): Participants treated with standard guideline-based care for 24 hours. Blood pressure treatment thresholds will be used according to standard practice parameters
- Interventional (Experimental): Autoregulation-guided blood pressure management for 24 hours. Blood pressure will be measured every four hours by arm cuff; however, in lieu of predetermined blood pressure treatment thresholds, an optimal mean arterial pressure (MAP) range will be chosen based on limits of autoregulation calculated in real-time for the previous four hours for each participant. Choice of medications and dosing will be left to the primary clinical obstetrics team.
  Interventions: Device: NIRS based personalized blood pressure management

INTERVENTIONS:
Device: NIRS based personalized blood pressure management — In lieu of predetermined blood pressure treatment thresholds, an optimal MAP range will be chosen based on limits of autoregulation calculated in real-time for the previous four hours for each participant. Choice of medications and dosing will be left to the primary clinical obstetrics team.
  Arms: Interventional

SUMMARY:
The purpose of this study is to test a new approach to blood pressure management in postpartum preeclampsia. There will be two groups of patients in this early stage single center trial. Both groups of study participants (observational and interventional) will be treated with standard blood pressure medications while undergoing continuous non-invasive blood pressure and near infrared spectroscopy (NIRS) monitoring for 24 hours. The interventional group will have personalized blood pressure targets according to results of NIRS monitoring which will be updated in real time.

DETAILED DESCRIPTION:
Maternal neurological complications are a leading cause of postpartum severe maternal morbidity and maternal mortality (SMM/MM). The lack of biomarkers to identify women at highest risk of these rare, but devastating postpartum complications, including stroke, seizures, and posterior reversible encephalopathy syndrome, has impeded efforts to prevent neurological SMM/MM.

Impaired cerebral autoregulation may be such a biomarker. Preliminary results using transcranial Doppler (TCD) based techniques to quantify cerebral autoregulation have demonstrated severely impaired cerebral autoregulation in the postpartum period in some women. However, TCD is operator dependent, and cannot be used for extended monitoring due to discomfort. In contrast, near-infrared spectroscopy (NIRS) is fully automated and can be continued for hours at the bedside. Identifying personalized blood pressure (BP) targets using NIRS has been shown to improve outcomes in acute stroke patients, another population with impaired cerebral autoregulation. However, this method has not been applied in postpartum women.

The investigators are applying this novel approach to the management of postpartum preeclampsia (PEC) in a single-center, Phase II clinical trial, PROMIS (PROtecting Maternal brains from Injury and Stroke).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or older, within 6 weeks postpartum after a pregnancy lasting at least 20 weeks.
* Admitted to the inpatient obstetrics unit for treatment of preeclampsia with one or both of the following severe features:

  1. measured systolic BP ≥160 mmHg and/or diastolic BP ≥110 mmHg on two or more occasions, 15 minutes apart OR
  2. severe headache refractory to standard over-the-counter medications (acetaminophen, ibuprofen)

Exclusion Criteria:

* Acute ischemic stroke
* Acute intracerebral or subarachnoid hemorrhage ·
* Eclamptic seizures
* Any other neurological complication requiring transfer to the neurological intensive care unit or stroke step-down unit
* Prior history of stroke, seizures, traumatic brain injury, brain surgery, encephalitis, or demyelinating brain disease
* History of Reynaud's syndrome (contraindication to finger plethysmography)
* Inability to understand and consent to the study

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2023-05-04 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Percentage of time mean arterial pressure (MAP) is in the target range | 24 hours
  The total time (in minutes) each participant had their mean arterial blood pressure (MAP) values within their computed limits of autoregulation will be measured. The primary outcome is the percentage of time the MAP is within the personalized limits of autoregulation.

SECONDARY OUTCOMES:
Number of participants with neurological symptoms | 24 hours
  Number of participants with neurological symptoms. Neurological symptoms defined as ≥8/10 headache pain or blurred vision.
Number of participants with physiological biomarker evidence of cerebral hypoperfusion | 24 hours
  Tissue oxygenation index (TOI) is defined as the ratio of oxygenated to total tissue hemoglobin as measured by NIRS. After initial securing of Foresight cerebral forehead oximetry adhesive stickers, baseline TOI will be recorded after two minutes of monitoring. Hypoperfusion will be defined as >13% decrease from baseline TOI.
Number of participants with physiological biomarker evidence of cerebral hyperperfusion | 24 hours
  Tissue oxygenation index (TOI) is defined as the ratio of oxygenated to total tissue hemoglobin as measured by NIRS. After initial securing of Foresight cerebral forehead oximetry adhesive stickers, baseline TOI will be recorded after two minutes of monitoring. Hyperperfusion will be defined as a >2% increase from baseline TOI.

CONTACTS AND LOCATIONS:
Overall Officials: Eliza Miller, MD, MS, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center / NewYork-Presbyterian Hospital (NYP), New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kirschner M, Woolcock Martinez H, Haghighi N, Booker WA, Marshall R, Bello NA, Petersen N, Miller EC. Increased Blood Pressure Variability is Associated with More Time Spent Outside Personalized Limits of Cerebral Autoregulation in Postpartum Preeclampsia. Neurocrit Care. 2025 Dec;43(3):853-863. doi: 10.1007/s12028-025-02316-y. Epub 2025 Jul 8. PMID 40629211